CLINICAL TRIAL: NCT04446104
Title: A Randomized Open-label Prophylaxis Trial Among Migrant Workers at High-risk of COVID-19 (DORM Trial)
Brief Title: A Preventive Treatment for Migrant Workers at High-risk of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/00561
Record Dates: First submitted 2020-05-11; First posted 2020-06-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Ivermectin; Zinc; Povidone-Iodine; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hydroxychloroquine (Experimental): Participants will receive hydroxychloroquine tablet 400mg loading dose, followed by 200mg daily for 42 days
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets
- Ivermectin (Experimental): Participants will receive ivermectin tablet 12mg single dose
  Interventions: Drug: Ivermectin 3mg Tab
- Zinc/ Vitamin C (Experimental): Participants will receive zinc tablet 80 mg/vitamin C 500mg daily for 42 days
  Interventions: Drug: Zinc
- Povidone-iodine throat spray (Experimental): Participants will receive povidone-iodine throat spray (3 times daily) for 42 days
  Interventions: Drug: Povidone-Iodine
- Vitamin C (Active Comparator): Participants will receive vitamin C tablet 500mg daily for 42 days
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets — Hydroxychloroquine tablet 400mg loading dose, followed by 200mg daily for 42 days
  Arms: Hydroxychloroquine
Drug: Ivermectin 3mg Tab — Ivermectin tablet 12mg single dose
  Arms: Ivermectin
Drug: Zinc — Zinc tablet 80 mg/vitamin C 500mg daily for 42 days
  Arms: Zinc/ Vitamin C
Drug: Povidone-Iodine — Povidone-iodine throat spray (3 times daily) for 42 days
  Arms: Povidone-iodine throat spray
Dietary Supplement: Vitamin C — Vitamin C tablet 500mg daily for 42 days
  Arms: Vitamin C

SUMMARY:
In December 2019, a novel coronavirus, now called COVID-19, emerged as a global health threat from Wuhan, China. Within weeks, the contagious virus spread within and between communities, causing a lower respiratory tract infection dominated by symptoms of fever, cough and sore throat. The incubation period was estimated at between 5 to 7 days, but could last as long as 14 days. Although COVID-19 causes a mostly mild and self-limiting disease, respiratory involvement has been reported in about 5% of the population, requiring supplemental oxygen and even ventilatory support to relieve hypoxia. Alveolar damage, fibrosis and consolidation have been reported in radiologic and post-mortem studies. Existing data suggest a mortality rate of COVID-19 is approximately 1-2%, higher among individuals with pre-existing comorbidities and in healthcare systems with suboptimal access to ventilatory support.

Given its high transmissibility, COVID-19 has quickly spread across the globe within a short interval. By 27 April 2020, over 3 million people around the world have been diagnosed with COVID-19, and more 200,000 have succumbed to the disease. As a proportion of patients manifest mild or no symptoms, these numbers are likely an underestimate of the actual number of patients with COVID-19. More disconcertingly, patients are known to shed viruses despite mild or no symptoms, making it essential that a collective approach against COVID-19 incorporate active pharmacological treatment to prevent or mitigate virus pathogenesis prior to its potential evolution to cause respiratory distress. To date, clinical trials have focused on the treatment of hospitalised patients diagnosed with COVID-19; only few have examined the clinical benefits of pharmacological agents despite few compelling in vitro data.

The relatively high transmission of COVID-19 in a closed dormitory environment of migrant workers in Singapore presents a real-life scenario where a prophylaxis treatment could reduce the impact of the disease. In Singapore, there are well grounded concerns an excess in cases could pose the possibility of strain in healthcare system and mentally drain her workers. The availability of an effective prophylaxis treatment is highly desirable to potentially reduce this burden. Data from the current study could also have implications on how future outbreaks in high-density areas should be managed, especially when residents are subjected to quarantine and isolation.

DETAILED DESCRIPTION:
This is a pragmatic, open-label, randomised study with 4 interventional and 1 control arms. Individuals will be recruited from migrant worker dormitories, and written informed consent taken prior to enrolment. Randomisation will be done by the level within the dormitory building and predetermined each day according to a randomisation schema done by an independent statistician. This will obviate the potential for bias due to drug exchange between study individuals.

The 5 arms consist of:

* Experimental arms

  1. Hydroxychloroquine tablet 400mg loading dose, followed by 200mg daily for 42 days (1,000 study subjects)
  2. Ivermectin tablet 12mg single dose (1,000 study subjects)
  3. Zinc tablet 80 mg/vitamin C 500mg daily for 42 days (1,000 study subjects)
  4. Povidone-iodine throat spray (3 times daily) for 42 days (1,000 study subjects)
* Control arm 5) Vitamin C tablet 500mg daily for 42 days (1,000 study subjects)

Study information sheet will be circulated in selected buildings within the dormitory 1-4 days before recruitment starts. All publicity materials and informed consent form will be translated to the different languages (e.g. Tamil, Bengali, Chinese, Burmese and Malay). A translator will be present to aid translation if necessary. Study subjects will be given ample time to ask questions relating to the study. Prospective participants will respond by showing up to recruitment stations at designated dates and times. Facilitators from the dormitory will be engaged to assist with the ground crowd-control. Prospective videos will be shown to inform the subject on the purpose, study inclusion and exclusion criteria, study medications, blood taking, reporting of adverse effects and follow-up visits. Informed consent will be taken before all study-related procedures are performed, including study eligibility. Translators will also help translate the daily questionnaires.

During the baseline recruitment,

1. History of symptoms, comorbidities and prior illnesses will be asked. Specific questions include presence or absence of the following symptoms: Fever, chills, myalgia, headache, diarrhoea, running nose, anosmia, loss of taste, sore throat, dry cough, shortness of breath.
2. Measurements of study subjects' parameters such as weight, height, temperature, pulse rate and blood pressure will be recorded. Subjects randomised to Ivermectin arm and subsequently found to weigh below 60 kg will be randomised to other treatment arms. Subjects randomised to hydroxychloroquine arm and found to have systolic blood pressure >150 mmHg and/or diastolic blood pressure >90 mmHg and/or heart rate >100 beats per minute will also be randomized to other treatment arms.
3. 12-lead electrocardiogram (ECG) will be performed in patients randomised to receive hydroxychloroquine. Only those with corrected QT values less than 450 ms, no cardiac arrhythmia and no ventricular hypertrophy will be allowed to receive hydroxychloroquine. Those with corrected QT values more than 450 ms, cardiac arrhythmia and ventricular hypertrophy will be randomised to other treatment arms.
4. Blood sample (20 mL) will be obtained to test Immunoglobulin G/M against SARS-CoV-2. Depending on the findings, additional tests will be performed to explore potential biological reasons underpinning these observations. The choice of markers may include pathway-specific biomarkers targeting inflammation, oxidative stress, lipid parameters, as well as organ-specific ones such as renal and liver parameters. Given the large sample size and high costs of analysis, the study team will prioritise more detailed investigations in a targeted group of patients depending on the final findings. None of these blood results is a screening criteria for study participation. The investigator will share abnormal to the study subjects abnormal results of their renal and liver parameters should these tests are tested following study completion. The extent on investigation, however, depends on funding support. In this study, renal and hepatic dysfunction will be based on physician-diagnosed and self-declaration on the part of the study subject. All clinical information will be verified by a senior physician on-site.
5. Study medications will be packed with clear instructions written on the packing bag. The package will be distributed to each subject based on the randomised treatment assigned.
6. Study participants will be given a study card to remind them to submit their symptoms daily and to record the times when they consume their medications. They will also be asked to present this card to doctors at the medical post or hospital should they seek medical assistance. In the events of acute respiratory infection and hospitalization, lab testing will be done as clinically indicated. Subjects on ventilator support who are not able to take oral medications may discontinue taking the study drug. However, subjects will remain in the study for collection of data on duration of mechanical ventilation for analysis.

During final study visit,

1. The study team, including investigators, will be present at the dormitory. A repeated blood sample (20mL) will be collected for serological tests. Measurements of study subjects' parameters such as weight (using Tanita BC-418 and Tanita BC-420MA for bio-electrical impedance analysis), height, blood pressure will be taken. ECG will be done only for subjects in hydroxychloroquine arm. History will be taken including symptoms of fever, chills, myalgia, headache, diarrhoea, running nose, anosmia, loss of taste, sore throat, dry cough, shortness of breath and the duration of such symptoms, if any.
2. Balance medication and packaging retrieval to do medication accounting and checking for adherence to assigned treatment arm
3. Discharged from study if no adverse events to follow-up.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the of following criteria to be included in this study:

* Men residing in dormitory aged 21-60 years
* Willing and able to give informed consent
* Able to understand instructions and consume study medications according to the study protocol.
* Weight more than 40kg
* Owns a mobile phone (with wireless fidelity and/or 3G connection and able to fill in online forms.

Exclusion Criteria:

Subjects who have any of the following criteria at baseline will be excluded from participating in this study:

* Symptoms of acute respiratory illness (e.g. fever, runny nose, sore throat, cough, breathlessness, loss of smell and loss of taste) for the past 30 days
* Known current or history of SARS-CoV-2 infection
* Unable to read English or any of the available local languages used for this clinical trial
* History of cardiac or neurological diseases
* History of retinal diseases
* History of diabetes on insulin treatment
* History of depression
* History of chronic alcohol use
* History of renal or hepatic dysfunction
* History of glucose-6-phosphate dehydrogenase deficiency
* History of anaemia, after exposure to any given medications
* History of thyroid disorder, hyperthyroidism, or sensitivity to iodine
* History of allergies with systemic presentation to any given medication (e.g.: swelling of the face, throat, eyes and lips, respiratory disturbances, asthmatic attacks, widespread skin blistering or urticaria (hives))
* Concomitant medication that may lead to cardiac arrhythmia (azithromycin, amitriptyline, cimetidine, citalopram, nortriptyline, pantoprazole, quetiapine etc).
* Unwilling to comply with study dosing, instructions or restrictions.

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4257 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed COVID-19 in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42

SECONDARY OUTCOMES:
Acute respiratory illness in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
  Acute respiratory illness is defined by acute onset with any key respiratory symptoms including cough, shortness of breath, sore throat, runny nose and change in smell.
Febrile respiratory illness in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Rate of hospitalization for COVID-19 and non-COVID-19 related indications in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Rate of oxygen supplementation and mechanical ventilation in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Duration of oxygen supplementation and mechanical ventilation in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Length of hospital stay in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Rate of laboratory-confirmed COVID-19 in treatment arms (hydroxychloroquine, ivermectin, zinc and povidone iodine) | At the end of study dosing, which is day 42
Adverse events and serious adverse events in control arm (Vitamin C) | At the end of study dosing, which is day 42
Drug discontinuation due to adverse events in control arm (Vitamin C) | At the end of study dosing, which is day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Tuas South Dormitory, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teng O, Quek AML, Ooi DSQ, Wang S, Fragata L, Ng IXQ, Cui J, Chen J, Hartman M, Hutchinson PE, Tambyah PA, Seet RCS. High CD4(+) T-cell responses in seronegative individuals following SARS-CoV-2 exposure during a dormitory outbreak. Int J Infect Dis. 2025 Oct;159:108024. doi: 10.1016/j.ijid.2025.108024. Epub 2025 Aug 20. PMID 40845939